CLINICAL TRIAL: NCT07376577
Title: A Randomized Controlled Trial on the Efficacy and Safety of Anricofen Combined With Ciprofol for Deep Sedation in Elderly Patients Undergoing Endoscopic Retrograde Cholangiopancreatography
Brief Title: Efficacy and Safety of Anricofen Combined With Ciprofol for Deep Sedation in Elderly Patients Undergoing ERCP
Acronym: Anricofen Cipr
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: The First Affiliated Hospital of Xinxiang Medical College (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: XYFY-IIT-ANES-ERCP-2025-01
Record Dates: First submitted 2026-01-16; First posted 2026-01-29 (Actual); Last update posted 2026-01-29 (Actual); Status verified 2026-01

CONDITIONS: Anesthesia; Sedation; ERCP; Ciprofol
MeSH Terms: interventions — Sufentanil; (2-(1R)-1-cyclopropyl)ethyl-6-isopropyl-phenol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Anricofen 0.3 μg/kg + Ciprofol 1.0 mg/kg (Experimental)
  Interventions: Drug: Anricofen; Drug: Ciprofol
- Anricofen 0.5 μg/kg + Ciprofol 1.0 mg/kg (Experimental)
  Interventions: Drug: Anricofen; Drug: Ciprofol
- Sufentanil 0.1 μg/kg + Ciprofol 1.0 mg/kg (Active Comparator): Participants receive intravenous sufentanil at a dose of 0.1 μg/kg (standard clinical dose) combined with ciprofol at 1.0 mg/kg for induction of deep sedation prior to ERCP. This regimen serves as the active control. Supplemental doses (one-third of the initial sufentanil dose and one-fourth of the initial ciprofol dose) may be administered during the procedure if needed based on behavioral pain score (BPS >3) or body movements.
  Interventions: Drug: Sufentanil; Drug: Anricofen

INTERVENTIONS:
Drug: Sufentanil — Sufentanil is a potent synthetic opioid analgesic acting primarily on μ-opioid receptors. It is commonly used for analgesia during surgical and endoscopic procedures. In this study, it serves as the active comparator in combination with ciprofol. It is administered intravenously.
  Arms: Sufentanil 0.1 μg/kg + Ciprofol 1.0 mg/kg
Drug: Anricofen — Anricofen is a novel peripherally selective κ-opioid receptor agonist. It provides analgesia primarily through peripheral mechanisms with minimal central nervous system penetration, thereby reducing the risk of respiratory depression and addiction compared to traditional μ-opioid agonists. It is administered intravenously.
Drug: Ciprofol — Ciprofol is a novel intravenous sedative agent with higher lipophilicity than propofol, leading to faster onset and recovery. It exhibits less cardiovascular depression compared to propofol and is suitable for procedural sedation, particularly in elderly patients. It is administered intravenously.
  Arms: Anricofen 0.3 μg/kg + Ciprofol 1.0 mg/kg; Anricofen 0.5 μg/kg + Ciprofol 1.0 mg/kg

SUMMARY:
Background: Endoscopic retrograde cholangiopancreatography (ERCP) is a key technique for treating pancreatobiliary diseases in the elderly. However, traditional sedative and analgesic regimens (e.g., sufentanil combined with propofol) are associated with a high incidence of respiratory depression, postoperative nausea and vomiting (PONV), and delayed recovery in elderly patients. Anricofen is a novel peripherally selective κ-opioid receptor agonist that provides analgesia with minimal central respiratory depression. Ciprofol is a new sedative agent characterized by rapid onset and quick recovery. The combination of these two drugs may offer a safer sedation and analgesia regimen for elderly patients undergoing ERCP.

Objective: To evaluate the efficacy and safety of anricofen combined with ciprofol for deep sedation in elderly patients undergoing ERCP, compared with the traditional regimen (sufentanil combined with ciprofol).

Methods: This is a single-center, randomized, double-blind, controlled trial. A total of 141 elderly patients aged 60-90 years with ASA physical status II-III scheduled for elective ERCP will be enrolled and randomly assigned in a 1:1:1 ratio to three groups: Anricofen 0.3 μg/kg + Ciprofol 1.0 mg/kg, Anricofen 0.5 μg/kg + Ciprofol 1.0 mg/kg, or Sufentanil 0.1 μg/kg + Ciprofol 1.0 mg/kg. The primary efficacy endpoint is the intraoperative pain control success rate (proportion of time with Behavioral Pain Scale [BPS] score ≤3 ≥90%). The primary safety endpoint is the incidence of respiratory depression (respiratory rate <10 breaths/min or SpO₂ <90% requiring intervention). Secondary outcomes include sedation depth, body movement episodes, recovery time, PONV incidence, and others.

Significance: This study aims to provide a sedation and analgesia regimen with lower risk of respiratory depression and faster recovery for elderly patients undergoing ERCP.

ELIGIBILITY:
Inclusion Criteria:

-

Inclusion Criteria:

1. Age 60-90 years.
2. American Society of Anesthesiologists (ASA) physical status II or III.
3. Scheduled for elective endoscopic retrograde cholangiopancreatography (ERCP).
4. Body mass index (BMI) between 18 and 30 kg/m².
5. Willing and able to provide written informed consent.

Exclusion Criteria:

1. Severe neurological disorders (acute stroke, uncontrolled seizures, epilepsy).
2. Psychiatric disorders or cognitive impairment (Mini-Mental State Examination score <24).
3. Uncontrolled hypertension (preoperative blood pressure ≥180/110 mmHg) or hypotension (<90/60 mmHg).
4. Severe cardiac disease: sinus bradycardia, sick sinus syndrome, unstable angina, or myocardial infarction within the past 3 months.
5. Severe hepatic or renal dysfunction.
6. Difficult airway or severe respiratory disease.
7. Achalasia.
8. Known allergy to anricofen, sufentanil, ciprofol, or other study medications.
9. Use of opioid analgesics or sedatives within 7 days prior to surgery.
10. Preoperative pulse oxygen saturation (SpO₂) <90% on room air.
11. Pregnancy or lactation.
12. Participation in any other drug clinical trial within the past 3 months.
13. Refusal to participate in the study.

Exclusion Criteria:

-

Ages: 60 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 141 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2028-03-01 (Estimated); Study Completion 2028-05-01 (Estimated)

PRIMARY OUTCOMES:
Intraoperative Pain Control Success Rate | During the ERCP procedure (from induction to end of procedure)

IPD SHARING:
Plan to Share IPD: Undecided